CLINICAL TRIAL: NCT04542148
Title: Glycemic Control After Antenatal Corticosteroids in Women With Pregestational and Gestational Diabetes (Close the GAP)
Brief Title: Glycemic Control After Antenatal Corticosteroids in Women With Pregestational and Gestational Diabetes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ashley N. Battarbee, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300005848
Record Dates: First submitted 2020-08-18; First posted 2020-09-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Preterm Birth; Pregnancy, High Risk; Diabetes, Gestational
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Premature Birth; Diabetes, Gestational | interventions — Insulin Aspart; Insulin Lispro; Insulin Glargine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Sliding Scale Insulin (Experimental): Addition of supplemental sliding scale insulin to home insulin regimen for maximum of 5 days after antenatal corticosteroids
  Interventions: Drug: Sliding Scale Insulin; Device: Dexcom G6 Professional Continuous Glucose Monitor
- Up-Titration of Home Insulin (Experimental): Increase in home insulin regimen based on standardized algorithm for maximum of 5 days after antenatal corticosteroids
  Interventions: Drug: Up-Titration of Home Insulin; Device: Dexcom G6 Professional Continuous Glucose Monitor
- Continuous Insulin Infusion (Experimental): Discontinuation of home insulin regimen and receipt of continuous insulin infusion for maximum of 5 days after antenatal corticosteroids
  Interventions: Drug: Continuous Insulin Infusion; Device: Dexcom G6 Professional Continuous Glucose Monitor

INTERVENTIONS:
Drug: Sliding Scale Insulin — After antenatal corticosteroid administration, women will continue to receive long- and short-acting subcutaneous insulin injections as prescribed at home. In addition, they will receive supplemental short-acting insulin using a sliding scale based on postprandial glucose values. Capillary blood glucose values will be measured with fingersticks 4 times daily (fasting and 1-hour postprandial).
  Other Names: Aspart; Lispro
  Arms: Sliding Scale Insulin
Drug: Up-Titration of Home Insulin — After antenatal corticosteroid administration, women will receive long- and short-acting subcutaneous insulin injections at increased dosages compared to that prescribed at home. Insulin will be increased by 30% on the day that they receive their 1st dose of antenatal corticosteroids (day 1), 50% on day 2, 50% on day 3, 30% on day 4, and 15% increase on day 5. On day 6 they will return to their home insulin regimen. Capillary blood glucose values will be measured with fingersticks 4 times daily (fasting and 1-hour postprandial).
  Other Names: Glargine; NPH; Aspart; Lispro; Regular insulin
  Arms: Up-Titration of Home Insulin
Drug: Continuous Insulin Infusion — After antenatal corticosteroid administration, women will discontinue their home insulin regimen and be placed on a continuous insulin infusion with insulin boluses and titration of infusion rate per institutional L&D protocol. Capillary blood glucose values will be measured with fingersticks every hour.
  Other Names: Regular insulin
  Arms: Continuous Insulin Infusion
Device: Dexcom G6 Professional Continuous Glucose Monitor — Masked Dexcom G6 Pro devices will be worn for 10 days.
  Other Names: G6 Pro

SUMMARY:
There is a fundamental gap in understanding the maternal and neonatal effects of antenatal corticosteroid (ACS) administration in women with threatened preterm birth (PTB) who have diabetes. Since the initial discovery of ACS for neonatal benefit in 1972, more than 40 randomized controlled trials have been performed evaluating its efficacy. However, none of these trials have included women with T2DM, and there is limited data among women with gestational diabetes. While ACS have been shown to reduce neonatal morbidity associated with PTB in non-diabetic women, the side effects of ACS (maternal hyperglycemia and fetal hyperinsulinemia) may mitigate the neonatal benefit of ACS in women with diabetes. Before neonatal benefit of ACS can be evaluated in this population, the first step is to optimize maternal glycemic control after ACS. Previous studies evaluating maternal hyperglycemia after ACS have been limited by small sample size, retrospective study design, or insufficient glucose data. Use of continuous glucose monitoring (CGM) in a randomized clinical trial provides a unique opportunity to overcome these challenges. Our long-term goal is to improve maternal and child health among women with diabetes as an independently funded clinical researcher. The research objectives of this proposal are to test the efficacy of three treatment strategies at achieving maternal glycemic control after ACS and evaluate the association between maternal glycemic control and neonatal outcomes. Our central hypothesis is that treatment with a continuous insulin infusion will improve maternal glycemic control, which is key to improving neonatal outcomes, but at the cost of less patient satisfaction and more health resource utilization. This hypothesis will be tested by pursuing the following specific aims: 1) Test the efficacy of three treatment strategies (addition of sliding scale insulin, up-titration of home insulin, and continuous insulin infusion) at achieving maternal glycemic control after ACS and 2) Quantify the association between maternal glycemic control after ACS and neonatal morbidity. Completion of these aims will determine the optimal strategy to achieve maternal glycemic control after ACS and inform a larger, multicenter trial to improve neonatal outcomes among women with diabetes and threatened PTB.

DETAILED DESCRIPTION:
Eligible, consenting women with medication-treated gestational or pregestational type 2 diabetes receiving ACS at 23 0/7 - 36 5/7 weeks' gestation for threatened PTB will be enrolled and randomized in a 1:1:1 ratio to receive 1) addition of sliding scale insulin to their home insulin regimen, 2) up-titration of their home insulin regimen, or 3) discontinuation of their home insulin regimen and initiation of a continuous insulin infusion. The randomization sequence will be created by the study statistician in a permuted block design, and assignments will be centrally allocated using the Research Electronic Data Capture (REDCap) application. Study investigators will be masked to the randomization sequence and varying block sizes.

Regardless of treatment group, all women will receive Dexcom G6 Professional CGM for 10 days. The device will be applied by research staff or if desired, by the patient herself, under direct supervision by research staff. The CGM sensor will be applied to the patient's abdomen away from skin folds, where there is hair, near the waistband or areas of scarring, tatoos, irritation or open wounds. An additional waterproof adhesive will be applied to help prevent the sensor from being dislodged and finally the transmitter will be attached. The patient will be provided a handout with instructions for care. The Professional CGM device will ensure both patients and providers are masked to CGM data, which will be used for research purposes only as CGM is not readily available to guide insulin titration in most clinical settings. Capillary blood glucose testing, the method routinely used in clinical practice, will be used to guide insulin titration for each treatment group. Women assigned to the sliding scale insulin group will continue their home insulin regimen and receive supplemental insulin as needed for post-prandial hyperglycemia based on capillary blood glucose testing 4 times daily (fasting and 1-hour post-prandial) for 5 days after ACS. Women assigned to the up-titration of home insulin group will have their home insulin dosages increased based on an algorithm with capillary blood glucose testing 4 times daily and additional sliding scale insulin as needed for post-prandial hyperglycemia. For example, if a woman's baseline insulin regimen includes a total of 70 units of daily insulin (NPH 30 units in the morning (qAM), NPH 10 units at bedtime (qPM), and Aspart 10 units with each meal), then on day 2 after ACS she will receive 50% more or 105 units total (NPH 45 units qAM, NPH 15 units qPM, and Aspart 15 units with each meal). Women assigned to the continuous insulin infusion group will have their home insulin discontinued and receive a continuous insulin infusion based on hourly capillary blood glucose testing for 5 days after ACS. Given the high acuity of insulin infusion management these women will be monitored on L&D, but women in the other two treatment groups may be managed on L&D or on the Antepartum unit at the discretion of the primary provider. Regardless of treatment group, all women will be allowed to eat as long as it is deemed safe by the primary provider. If women assigned to receive the sliding scale insulin group or the up-titration of home insulin group are made nil per os (NPO) at any time after enrollment, they will be placed on the continuous insulin infusion per protocol with hourly capillary blood glucose testing. Once a diet is resumed, they will be switched back to the insulin algorithm.

Upon completion of the study intervention, all women will complete the Diabetes Treatment Satisfaction Questionnaire (DTSQ) to assess satisfaction with their insulin treatment strategy. The DTSQ is one of the most widely used treatment questionnaires as it is internationally validated and approved by the World Health Organization and International Diabetes Federation and available in over 100 different languages. The questionnaire is composed of 8 questions, each of which are scored on a scale ranging from 0 ("very dissatisfied or inconvenient") to 6 ("very satisfied or convenient"). The first section assesses treatment satisfaction and includes 6 questions that ask about 1) satisfaction with treatment, 2) flexibility, 3) convenience, 4) understanding of diabetes, 5) recommend treatment to others, and 6) willingness to continue. The second section consists of 2 questions that assess the burden of hyper- and hypoglycemia. Overall treatment satisfaction is measured by the sum of the scores on the first 6 questions, and a higher score indicates higher satisfaction (maximum score of 36). The DTSQ is particularly well-suited for use in this study because it is able assess treatment satisfaction regardless of the specific treatment method, and it is easy to answer without placing a large burden on patients.

Other than glycemic management during the 5 days after ACS, antenatal care (fetal testing, maternal laboratory evaluation, timing and mode of delivery) will be at the discretion of the primary obstetric provider. Umbilical cord blood will be collected at delivery and stored at the University of Alabama at Birmingham (UAB) for analysis at the conclusion of the trial. After birth, all neonates born to women with diabetes have a heelstick performed to measure capillary blood glucose as part of standard of care. Additional neonatal care after birth will be at the discretion of the primary neonatal provider.

Comprehensive baseline maternal data and maternal and neonatal outcomes will be abstracted from the UAB electronic medical record and Professional CGM devices. Additionally, measures of health resource utilization will be collected such as duration of time on labor and delivery, number of capillary blood glucose tests, treatments administered such as insulin, intravenous fluids, and dextrose for hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Gestational or pregestational type 2 diabetes mellitus treated with daily insulin injection(s) or oral hypoglycemic agents such as metformin
* Hospitalized for antenatal corticosteroid administration in anticipation of preterm birth
* Gestational age 23 0/7 weeks - 36 5/7 weeks
* Maternal age 18-50

Exclusion Criteria:

* Planned delivery < 72 hours after 1st dose of antenatal corticosteroids
* More than 16 hours after 1st dose of antenatal corticosteroids
* Major fetal anomaly
* Triplet or higher order multiple gestation

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The primary aim of the study is an intervention unique to pregnancy. Male and female neonates will be included.
Enrollment: 120 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time In Range | During study intervention assessed for maximum of 5 days after ACS
  Percent time glucose in range (65-140mg/dL) on CGM

SECONDARY OUTCOMES:
Time Above Range | During study intervention assessed for maximum of 5 days after ACS
  Percent time glucose above range (>140mg/dL) on CGM
Time Below Range | During study intervention assessed for maximum of 5 days after ACS
  Percent time glucose below range (<65mg/dL) on CGM
Additional insulin requirement | During study intervention assessed for maximum of 5 days after ACS
  Percent increase in daily insulin requirements compared to home regimen
Glucose variability | During study intervention assessed for maximum of 5 days after ACS
  Coefficient of variation (glucose standard deviation / mean glucose) on CGM
Patient satisfaction | Upon completion of study intervention, on average 5 days after enrollment
  Score on modified Diabetes Treatment Satisfaction Questionnaire (questions 1, 4, 5, 6, 7, 8) with score range from 0-36 with 0 being not satisfied and 36 being very satisfied
Neonatal composite respiratory morbidity | Birth to hospital discharge, assessed up to 28 days
  Composite including need for continuous positive airway pressure or high-flow nasal cannula of >=0.30 for >=12 continuous hours, respiratory distress syndrome, or mechanical ventilation
Initial neonatal glucose | Birth to 2 hours of life
  Initial capillary neonatal glucose in mg/dL measured by heelstick
Umbilical cord blood C-peptide | Delivery
  C-peptide concentration (mcg/L) in the umbilical cord blood as measure of fetal insulin status
Umbilical cord blood insulin | Delivery
  Insulin concentration (mcg/L) in the umbilical cord blood as measure of fetal insulin status
Umbilical cord blood cortisol | Delivery
  Cortisol concentration (mcg/L) in the umbilical cord blood as measure of fetal HPA axis
Umbilical cord blood surfactant protein A (SP-A) | Delivery
  Fetal surfactant protein A
Umbilical cord blood surfactant protein B (SP-B) | Delivery
  Fetal surfactant protein B
Umbilical cord blood surfactant protein C (SP-C) | Delivery
  Fetal surfactant protein C
Umbilical cord blood surfactant protein D (SP-D) | Delivery
  Fetal surfactant protein D

CONTACTS AND LOCATIONS:
Overall Officials: Ashley N Battarbee, MD, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Oregon Health and Science University, Portland, Oregon
  - University of South Carolina Greenville / Prisma Health-Upstate, Greenville, South Carolina
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Rowley WR, Bezold C, Arikan Y, Byrne E, Krohe S. Diabetes 2030: Insights from Yesterday, Today, and Future Trends. Popul Health Manag. 2017 Feb;20(1):6-12. doi: 10.1089/pop.2015.0181. Epub 2016 Apr 28. PMID 27124621
- [Background] Boyle JP, Thompson TJ, Gregg EW, Barker LE, Williamson DF. Projection of the year 2050 burden of diabetes in the US adult population: dynamic modeling of incidence, mortality, and prediabetes prevalence. Popul Health Metr. 2010 Oct 22;8:29. doi: 10.1186/1478-7954-8-29. PMID 20969750
- [Background] Crowley PA. Antenatal corticosteroid therapy: a meta-analysis of the randomized trials, 1972 to 1994. Am J Obstet Gynecol. 1995 Jul;173(1):322-35. doi: 10.1016/0002-9378(95)90222-8. No abstract available. PMID 7631713
- [Background] Roberts D, Brown J, Medley N, Dalziel SR. Antenatal corticosteroids for accelerating fetal lung maturation for women at risk of preterm birth. Cochrane Database Syst Rev. 2017 Mar 21;3(3):CD004454. doi: 10.1002/14651858.CD004454.pub3. PMID 28321847
- [Background] Amiya RM, Mlunde LB, Ota E, Swa T, Oladapo OT, Mori R. Antenatal Corticosteroids for Reducing Adverse Maternal and Child Outcomes in Special Populations of Women at Risk of Imminent Preterm Birth: A Systematic Review and Meta-Analysis. PLoS One. 2016 Feb 3;11(2):e0147604. doi: 10.1371/journal.pone.0147604. eCollection 2016. PMID 26841022
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 171: Management of Preterm Labor. Obstet Gynecol. 2016 Oct;128(4):e155-64. doi: 10.1097/AOG.0000000000001711. PMID 27661654
- [Background] Battarbee AN, Aliaga S, Boggess KA. Management of diabetic women with threatened preterm birth: a survey of Maternal-Fetal Medicine providers. J Matern Fetal Neonatal Med. 2020 Sep;33(17):2941-2949. doi: 10.1080/14767058.2019.1566307. Epub 2019 Jan 24. PMID 30678514
- [Background] Ramirez-Torres MA, Perez-Monter SE, Espino y Sosa S, Ibarguengoitia-Ochoa F. [Effect of betamethasone in blood glucose levels in pregnant diabetic women at risk of preterm birth]. Ginecol Obstet Mex. 2011 Sep;79(9):565-71. Spanish. PMID 21966858
- [Background] Mathiesen ER, Christensen AB, Hellmuth E, Hornnes P, Stage E, Damm P. Insulin dose during glucocorticoid treatment for fetal lung maturation in diabetic pregnancy: test of an algorithm [correction of analgoritm]. Acta Obstet Gynecol Scand. 2002 Sep;81(9):835-9. doi: 10.1034/j.1600-0412.2002.810906.x. PMID 12225298
- [Background] Kaushal K, Gibson JM, Railton A, Hounsome B, New JP, Young RJ. A protocol for improved glycaemic control following corticosteroid therapy in diabetic pregnancies. Diabet Med. 2003 Jan;20(1):73-5. doi: 10.1046/j.1464-5491.2003.00853.x. PMID 12519324
- [Background] Refuerzo JS, Garg A, Rech B, Ramin SM, Vidaeff A, Blackwell SC. Continuous glucose monitoring in diabetic women following antenatal corticosteroid therapy: a pilot study. Am J Perinatol. 2012 May;29(5):335-8. doi: 10.1055/s-0031-1295642. Epub 2011 Nov 17. PMID 22094918
- [Background] Battarbee AN, Anderson SB, Tita ATN, Harper LM. Methods of Glycemic Control and Neonatal Outcomes after Antenatal Corticosteroid Administration among Women with Pregestational Diabetes. Am J Perinatol. 2020 Nov;37(13):1351-1356. doi: 10.1055/s-0039-1693717. Epub 2019 Jul 31. PMID 31365928
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 201: Pregestational Diabetes Mellitus. Obstet Gynecol. 2018 Dec;132(6):e228-e248. doi: 10.1097/AOG.0000000000002960. PMID 30461693
- [Background] International Association of Diabetes and Pregnancy Study Groups Consensus Panel; Metzger BE, Gabbe SG, Persson B, Buchanan TA, Catalano PA, Damm P, Dyer AR, Leiva Ad, Hod M, Kitzmiler JL, Lowe LP, McIntyre HD, Oats JJ, Omori Y, Schmidt MI. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Diabetes Care. 2010 Mar;33(3):676-82. doi: 10.2337/dc09-1848. No abstract available. PMID 20190296
- [Background] Miracle X, Di Renzo GC, Stark A, Fanaroff A, Carbonell-Estrany X, Saling E; Coordinators Of World Associatin of Perinatal Medicine Prematurity Working Group. Guideline for the use of antenatal corticosteroids for fetal maturation. J Perinat Med. 2008;36(3):191-6. doi: 10.1515/JPM.2008.032. PMID 18576926
- [Background] Feig DS, Donovan LE, Corcoy R, Murphy KE, Amiel SA, Hunt KF, Asztalos E, Barrett JFR, Sanchez JJ, de Leiva A, Hod M, Jovanovic L, Keely E, McManus R, Hutton EK, Meek CL, Stewart ZA, Wysocki T, O'Brien R, Ruedy K, Kollman C, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. Continuous glucose monitoring in pregnant women with type 1 diabetes (CONCEPTT): a multicentre international randomised controlled trial. Lancet. 2017 Nov 25;390(10110):2347-2359. doi: 10.1016/S0140-6736(17)32400-5. Epub 2017 Sep 15. PMID 28923465
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Piper JM, Langer O. Does maternal diabetes delay fetal pulmonary maturity? Am J Obstet Gynecol. 1993 Mar;168(3 Pt 1):783-6. doi: 10.1016/s0002-9378(12)90819-4. PMID 8456880
- [Background] Piper JM, Xenakis EM, Langer O. Delayed appearance of pulmonary maturation markers is associated with poor glucose control in diabetic pregnancies. J Matern Fetal Med. 1998 May-Jun;7(3):148-53. doi: 10.1002/(SICI)1520-6661(199805/06)7:33.0.CO;2-K. PMID 9642613
- [Background] Saisho Y. Use of Diabetes Treatment Satisfaction Questionnaire in Diabetes Care: Importance of Patient-Reported Outcomes. Int J Environ Res Public Health. 2018 May 9;15(5):947. doi: 10.3390/ijerph15050947. PMID 29747423